CLINICAL TRIAL: NCT03297866
Title: Effectiveness of Different Incentive Models in Booster up the Second Follow up Response Rate
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Other Study IDs: Incentive schemes 2017
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: To Test the Effectiveness of Different Incentive Models for Increasing the Follow-up Response Rate in the Current Smoker Subject

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Incentive schemes 1: No incentive will be given after completing the follow-up survey
- Incentive schemes 2: Receiving $100 supermarket coupon after completing the follow-up survey
- Incentive schemes 3: Receiving $200 supermarket coupon after completing the follow-up survey
- Incentive schemes 4: Receiving $100 supermarket coupon before completing the follow-up survey and another $100 supermarket coupon after completing the follow-up survey

SUMMARY:
Aim to test the effectiveness of different incentive models for increasing the follow-up response rate in the current smoker subject.

DETAILED DESCRIPTION:
According to the Hong Kong Census and Statistic Department, 10.5% of the Hong Kong population who aged 15 years or above are daily smokers (Thematic Household Survey Report - Report No. 59, 2016). The smoking prevalence was estimated from a thematic household survey that has been conducted every 2 or 3 years. Another population-based survey related to tobacco control is the Tobacco Control Policy-related Survey conducted by the Hong Kong Council on Smoking and Health and the University of Hong Kong. Both surveys were in a cross-sectional design and no follow-up was done. A cohort study with follow-up data could provide more insights for the causal relationship. However, most people are not willing to complete follow-up survey and the response rate is often low (Mellahi, 2016). The low survey response rate could lead to statistically bias in the research funding (Pit, 2014). Therefore, cohort surveys need to provide attractive monetary incentive to the interviewee to increase the response rate (Pit, 2014).

This study aims to assess and compare the 3-month response rate of a follow-up survey due to different financial incentive schemes. The findings will be used for a feasibility assessment of future cohort studies of evaluating tobacco control measures and public opinion, and exploration of appropriate incentive scheme.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 or above
* Cantonese or Mandarin speakers

Exclusion Criteria:

* Unable to provide a consent form
* Speak language other than Cantonese and Mandarin

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Hong Kong residents
Sampling Method: Probability Sample
Enrollment: 1246 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Proportion of respondents who will complete the 3-month follow-up | Finish all telephone survey by Jan 2018
  Proportion of respondents who will complete the 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Public Opinion Programme, the University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Cheung YTD, Weng X, Wang MP, Ho SY, Kwong ACS, Lai VWY, Lam TH. Effect of prepaid and promised financial incentive on follow-up survey response in cigarette smokers: a randomized controlled trial. BMC Med Res Methodol. 2019 Jul 4;19(1):138. doi: 10.1186/s12874-019-0786-9. PMID 31272393